CLINICAL TRIAL: NCT02767765
Title: Pilot Study for Evaluating the Efficacy and Tolerability of Induction Therapy With Recombinant Human Erythropoietin Beta (rHuEPO) NeoRecormon® - at High Dose in Anemic Cancer Patients Treated With Chemotherapy
Brief Title: A Study of Recombinant Human Erythropoietin Beta (NeoRecormon) in Anemic Cancer Participants Treated With Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17435
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Erythropoietin; epoetin beta

ARMS (1):
- r-HuEPO (Experimental): Anemic cancer participants will receive r-HuEPO for 4 weeks.
  Interventions: Drug: r-HuEPO

INTERVENTIONS:
Drug: r-HuEPO — All participants will receive r-HuEPO for 4 weeks, at a dose of 10000 international units per day (IU/day) according to 6 days/week schedule for first 2 weeks and at a dose of 10000 IU/day according to 3 days/week schedule (participants with response to treatment at end of Week 2) or according to 6 days/week schedule (participants without response to treatment at end of Week 2) for next 2 weeks.
  Other Names: NeoRecormon

SUMMARY:
This study will evaluate the efficacy and tolerability of subcutaneous (SC) or intramuscular (IM) recombinant human erythropoietin beta (r-HuEPO) in participants with anemia and histologically or cytologically confirmed cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed cancer
* Participants who are treated with at least first line chemotherapy
* Hemoglobin less than (<) 11 grams per deciliter (g/dL)
* Participants able to receive iron supplement, if necessary

Exclusion Criteria:

* History of hypersensitivity to active or inactive excipients of r-HuEPO
* Insufficient controllable hypertension
* Thalassemic syndromes
* Anemia caused by hematic loss
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Italy (6):
  - Bari
  - Benevento
  - Cagliari
  - Campobasso
  - Napoli
  - Palermo

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Erythropoietin Beta (r-HuEPO): Anemic cancer participants received r-HuEPO (NeoRecormon) as subcutaneous (SC) or intramuscular (IM) injection for 4 weeks, at a dose of 10000 international units per day (IU/day) according to 6 days/week schedule for first 2 weeks and at a dose of 10000 IU/day according to 3 days/week schedule (participants with response to treatment at end of Week 2) or according to 6 days/week schedule (participants without response to treatment at end of Week 2) for next 2 weeks.
Period: Overall Study
Arm/Group | Recombinant Human Erythropoietin Beta (r-HuEPO)
Started | 61
Completed | 50
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Insufficient response | 1
Not completed — Lost to Follow-up | 2
Not completed — Investigator decision | 1
Not completed — Non-Compliance | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who received at least one dose of study medication.
Groups:
- r-HuEPO: Anemic cancer participants received r-HuEPO as SC or IM injection for 4 weeks, at a dose of 10000 IU/day according to 6 days/week schedule for first 2 weeks and at a dose of 10000 IU/day according to 3 days/week schedule (participants with response to treatment at end of Week 2) or according to 6 days/week schedule (participants without response to treatment at end of Week 2) for next 2 weeks.
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.31 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment
Description: Response to treatment was defined as an increase of greater than (>) 1 gram per deciliter (g/dL) in hemoglobin level (irrespective of the need of transfusion) from Baseline value at Week 4.
Time Frame: Week 4
Population: The intent-to-treat (ITT) analysis population included all enrolled participants who received study medication for at least 2 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
percentage of participants | 50.8

2. Secondary Outcome: Time to Response
Description: Time to response was defined as the time between the start of treatment and the increase in hemoglobin level >1 g/dL compared to baseline hemoglobin level. Time to response was estimated using Kaplan Meier method.
Time Frame: Baseline up to Week 4
Population: ITT analysis population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
days | 19 [15 to 36]

3. Secondary Outcome: Percentage of Participants With Response to Treatment After 2 Weeks of Study Treatment
Description: Response to treatment after 2 weeks of treatment was defined as presence of any of the following criteria: reticulocytes >40000 per microliter or >25% increase in soluble transferrin receptor or >0.5 g/dL increase in hemoglobin level.
Time Frame: Week 2
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
percentage of participants | 78.7

4. Secondary Outcome: Percentage of Participants With No Response to Treatment After 4 Weeks of Study Treatment
Description: "No Response" to treatment after 4 weeks was defined as meeting any of the following criteria: <1 g/dL increase in hemoglobin level or hemoglobin level <8.5 g/dL or need of transfusion. If a participant had an increase in hemoglobin level of >1 g/dL but required transfusion then the participant is considered as Non- Responder.
Time Frame: Week 4
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
percentage of participants | 50.8

5. Secondary Outcome: Percentage of Participants Who Required Transfusion
Time Frame: Baseline, Week 2, Week 4
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | r-HuEPO
Number analyzed (Participants) | 61
percentage of participants
  Baseline | 8.2
  Week 2 | 4.9
  Week 4 | 1.7

6. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) Questionnaire Score at Week 4
Description: FACT-An comprises of 4 subscales of 27-item (FACT-General scale [FACT-G]): physical well-being, social/family well-being, emotion well-being, functional well-being, and an additional concerns anemia subscale. All questions are rated on a scale from 0 to 4, where higher scores indicate more impact on quality of life. The physical well-being subscale consists of 7 questions with score range from 0-28; social/family well-being subscale consists of 7 questions with score range from 0-28; emotion well-being subscale consists of 6 questions with score range from 0-24; functional well-being subscale consists of 7 questions with score range from 0-28; anemia subscale consist of 20 questions with score range from 0-80. Total FACT-An score ranges from 0-188.
Time Frame: Baseline, Week 4
Population: All enrolled participants who completed the questionnaire at baseline were included in the analysis. Here, "n" represents number of participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | r-HuEPO
Number analyzed (Participants) | 56
units on a scale
  Baseline (n=56) | 23.59 (10.80)
  Change at Week 4 (n=35) | -6.23 (8.11)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 4
Description: Safety population
Arm/Group | r-HuEPO
Serious Adverse Events (participants affected / at risk) | 3/61
Other Adverse Events (participants affected / at risk) | 12/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | r-HuEPO (N=61)
Cachexia (Metabolism and nutrition disorders) | 1
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Presyncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | r-HuEPO (N=61)
Anaemia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Oedema peripheral (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Presyncope (Nervous system disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.